CLINICAL TRIAL: NCT00593125
Title: Levetiracetam (Keppra) Tolerability and Efficacy in Cocaine Abusing Methadone-maintained Patients.
Brief Title: Levetiracetam (Keppra) Tolerability in Cocaine Abusing Methadone-maintained Patients.
Acronym: Keppra
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Gerardo Gonzalez, MD, Yale University
Organization: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Yale-0508000534; UBC,Inc; VA HSS GG 0004
Record Dates: First submitted 2007-12-31; First posted 2008-01-14 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-09

CONDITIONS: Cocaine Dependence; Opioid Dependence
Keywords: cocaine; opioids; heroin; levetiracetam
MeSH Terms: conditions — Cocaine-Related Disorders; Opioid-Related Disorders | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): levetiracetam
  Interventions: Drug: levetiracetam

INTERVENTIONS:
Drug: levetiracetam — The participants will start receiving Levetiracetam 500mg in the mornings of the first day on week 2. The dose will be titrated every third day, until the target dose of 3000mg/day is achieved by week 4. The study medication must be titrated to 3000 mg/day or to the subject's maximum tolerated dose (MTD). The physician overseeing this titration as well as all study staff will not be blind to the subject's medication administration. The medication will be discontinued over a two-week period
  Other Names: Keppra

SUMMARY:
The proposed investigation will use methadone maintained patients who have concurrent cocaine dependence in order to take advantage of the excellent (over 80%) treatment retention in this patient group and to maximize treatment compliance by daily observed medication with both methadone and levetiracetam. In the initial patients we will explore the tolerability of escalating doses of levetiracetam as well as its potential role in reducing cocaine use, as monitored by self-report and verified by three-times weekly urine toxicology testing in methadone treated patients.The specific aim of this study is to evaluate the tolerability and efficacy of levetiracetam 3 grams/day in modifying cocaine-using behavior, reducing cocaine craving and attenuating cocaine's reinforcing effect among methadone-maintained patients

DETAILED DESCRIPTION:
This 12-week open-label clinical trial will provide treatment for 15 cocaine-dependent opioid dependent patients. Participants, aged 18-65 years, will receive levetiracetam 3000 mg/day while concurrently receiving treatment with methadone. Baseline cocaine use will be determined during the first week of treatment participation.

The study design will have three overlapping phases that are summarized below: 1) A one week methadone fixed induction (week 1) and flexible stabilization phase (weeks 2-9); 2) an 8-week "treatment" phase (weeks 2-9), consisting of slow titration and stabilization on study medication; and 3) a four week "taper, detoxification or transfer" phase (weeks 9-12).

During the first week of induction onto methadone, participants will be administered fixed increasing doses of methadone starting at 30 mg daily and increased to 60 mg daily by the end of the first week. This methadone dose will be adjusted for stabilization of opiate withdrawal symptoms using a flexible dosing from 40 mg up to 150 mg. This range has been found to be adequate for the vast majority of patients receiving methadone in our program and is designed to accommodate participants who may not be able to tolerate the higher maintenance doses or may still experience withdrawal symptoms, respectively. We may increase or decrease this amount on a case-by-case basis based on physician assessment of self-reported and observed symptoms.

Starting on week 2 subjects will receive levetiracetam 500mg/day and this dose will be slowly titrated to a total of 3000mg/day or maximum tolerated dose (MTD). Subjects will remain on their full dosage through week 8.

At the end of week 8, participants will undergo detoxification from methadone over a 4-week period (weeks 8-12) and discontinuation from levetiracetam over a concurrent 2-week period. All participants will receive weekly 1-hour of individual psychotherapy (Cognitive Behavioral Treatment) with experienced clinicians specifically trained to deliver the therapy and who will receive ongoing supervision. The primary outcomes will be reported medication side effects (medication tolerability), and reduction in cocaine use, as assessed by self-report and thrice-weekly urinalyses. Secondary outcomes will include weeks in treatment (retention), and change in measures of: cocaine craving, anxiety symptoms and opiate withdrawal symptoms. This study will occur at the Outpatient Treatment Research Program in Building 36 at the VA CT Healthcare System.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 18-65 years.
2. Participants must demonstrate current opioid dependence as determined by study physician, self-reported history of opioid dependence for one year and a positive urine of opiates. Participants may be transferred from other methadone maintenance programs, including the WHVA methadone program.
3. Participants also must be current users of cocaine with self-reported use of cocaine > 1 time/week in at least one month preceding study entry, cocaine-positive urine screen and score over 3 as assessed with the Severity Dependence Scale (Kaye & Darke 2002).
4. Women of childbearing age are eligible to be included in the study if they have a negative pregnancy test at screening, agree to adequate contraception to prevent pregnancy, to have monthly pregnancy tests, and they understand the risk of fetal toxicity due to medication and cocaine.

Exclusion Criteria:

1. Current diagnosis of other drug or alcohol dependence (other than opiates, cocaine or tobacco).
2. Patients with serious medical illness (e.g., major cardiovascular, renal, endocrine, hepatic, and serious neurological disorders including any history of seizures).
3. Patients with current serious psychiatric illness or history of psychosis, schizophrenia, bipolar type I disorder and subjects with suicidal or homicidal thoughts or taking psychotropic medications.
4. Women who are pregnant, nursing or refuse to use a reliable form of birth control or refuse monthly testing.
5. Screening liver function tests (SGOT or SGPT) greater than 3 times normal and renal function test (creatinine) greater than 1.5 mg/dl.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-01; Primary Completion 2007-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Medication emergent side-effects | 12-weeks

SECONDARY OUTCOMES:
Thrice weekly urine toxicology | 12 weeks
Weekly self-report of cocaine and opioid use | 12-weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gerardo Gonzalez, MD, Principal Investigator — Yale University
Locations (1):
- VA CT Healthcare System, West Haven, Connecticut, United States